CLINICAL TRIAL: NCT03803527
Title: Metabolomic Profiling of Eosinophilic Esophagitis Patients With Dysphagia for Biomarker Discovery
Brief Title: Metabolomic Profiling of Eosinophilic Esophagitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study did not receive the grant that was applied for to conduct the study.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-0074
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EST (Experimental): All subjects enrolled into the study will:
  * Complete a clinical history
  * Have vitals obtained
  * Complete Patient-reported outcomes
  * Have Esophageal mucosal biopsies collected as part of standard of care at the time of the most recent endoscopy to report the peak eosinophilia per hpf.
  * Complete the Esophageal String test
  Interventions: Procedure: Esophageal String Test

INTERVENTIONS:
Procedure: Esophageal String Test — An EST will be performed for a 1hour sampling period on the same day as the scheduled clinic visit. Subjects will be asked to swallow a capsule and the attached EST string will be taped to the cheek with tegaderm tape. At the completion of the 1-hour sampling period, the EST will be removed and it will immediately be processed and cryopreserved for metabolomics profiling.

SUMMARY:
A prospective longitudinal, observational study of adolescent and adults that will identify novel metabolites associated with dysphagia in Eosinophilic Esophagitis (EoE).

DETAILED DESCRIPTION:
In this study, the investigators seek to understand whether a metabolomic profile obtained from esophageal samples correlate with the symptom of dysphagia in adolescent and adults. The investigators hypothesize that intraluminal secreted metabolite(s) will change during episodes of dysphagia. The aim of the study will be to use a novel method of producing esophageal luminal samples, the esophageal string test, to capture esophageal metabolites when a patient is and is not experiencing dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Eosinophilic Esophagitis (EoE) and seen either at Children's Hospital Colorado or University of Colorado Hospital for scheduled outpatient clinical assessment or upper GI endoscopy

Exclusion Criteria:

* Acute food impaction at time of study
* Recent (within 2 months) use of systemic steroids
* Other known esophageal disease or esophageal injury (e.g. tracheoesophageal fistula, congenital stricture, caustic injury)
* known other inflammatory bowel disease
* inability to swallow the EST

Ages: 11 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Brief Esophageal Dysphagia Questionnaire | Time of Endoscopic Procedure
  Positive Dysphagia symptoms Measured by Brief Esophageal Dysphagia Questionnaire. The questionnaire asks questions about dysphagia symptoms and the scale is from 0 (rarely/never) to 5 (several times per day).

IPD SHARING:
Plan to Share IPD: No